CLINICAL TRIAL: NCT00892892
Title: Role of the Sympathetic Nerve System for the Pathogenesis and Progression of Chronic Kidney Failure
Brief Title: Sympathetic Nerve Activity in Renal Failure
Acronym: SNS in CRF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Re-No. 3186
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: sympatholytic treatment; sympathetic nerve activity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Rilmenidine; Nitrendipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Rilmenidine as a sympatholytic agent for three months
  Interventions: Drug: Rilmenidine
- Arm 2 (Active Comparator): Nitrendipine as a non-sympatholytic agent for three months
  Interventions: Drug: Nitrendipine

INTERVENTIONS:
Drug: Rilmenidine — 1 mg Rilmenidine per day versus
  Other Names: Hyperium
  Arms: Arm 1
Drug: Nitrendipine — 20 mg Nitrendipine per day
  Other Names: Bayotensin
  Arms: Arm 2

SUMMARY:
The primary purpose is to assess the role of sympathetic activation for the development and progression of chronic renal failure. Using microneurography sympathetic activity will be registered in various stages of kidney affection or failure and hypertension.

A sympatholytic agent will be compared with a non-sympatholytic drug to asses the effect sympathetic activation and on the progression of kidney disease.

The effects of a sympatholytic agent on cardiovascular reactivity to various stressors wil be examined.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure stages I-IV

Exclusion Criteria:

* pregnancy and lactation
* severe heart failure or ischemic heart disease
* patients with NYHA III-IV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
sympathetic activation for the development and progression of chronic renal failure | 3 months

SECONDARY OUTCOMES:
effects of a sympatholytic agent on cardiovascular reactivity to various stressors | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nurnberg
Locations (1):
- University of Erlangen-Nuremberg, CRC, med. Clinic 4, Erlangen, Bavaria, Germany